CLINICAL TRIAL: NCT00079105
Title: A Phase II Study VEPEMB In Patients With Hodgkin's Lymphoma Aged ≥ 60 Years; Vinblastine, Cyclophosphamide, Procarbazine, Prednisolone, Etoposide, Mitoxantrone, and Bleomycin in Treating Older Patients With Hodgkin's Lymphoma
Brief Title: A Phase II Study VEPEMB In Patients With Hodgkin's Lymphoma Aged ≥ 60 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000354225; UON-SHIELD (Other: Sponsor); EU-20346 (Other: Sponsor)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Cyclophosphamide; Etoposide; etoposide phosphate; Mitoxantrone; Prednisolone; Methylprednisolone; prednisolone phosphate; Procarbazine; Vinblastine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Treatment with VEPEMB - Vinblastine sulfate, Cyclophosphamide, Procarbazine hydrochloride, Prednisolone, Etoposide, Mitoxantrone hydrochloride, and Bleomycin sulfate
  Interventions: Biological: bleomycin sulfate; Drug: cyclophosphamide; Drug: etoposide; Drug: mitoxantrone hydrochloride; Drug: prednisolone; Drug: procarbazine hydrochloride; Drug: vinblastine sulfate
- Registration (No Intervention): Registration, without treatment

INTERVENTIONS:
Biological: bleomycin sulfate — Treatment
  Other Names: Blenoxane
  Arms: Treatment
Drug: cyclophosphamide — Treatment
  Other Names: Cytoxan
  Arms: Treatment
Drug: etoposide — Treatment
  Other Names: Eposin; Etopophos; Vepesid
  Arms: Treatment
Drug: mitoxantrone hydrochloride — Treatment
  Other Names: Novantrone
  Arms: Treatment
Drug: prednisolone — Treatment
  Other Names: Flo-Pred; Pediapred; Orapred
  Arms: Treatment
Drug: procarbazine hydrochloride — Treatment
  Other Names: Matulane
  Arms: Treatment
Drug: vinblastine sulfate — Treatment
  Other Names: Vincristine
  Arms: Treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinblastine, cyclophosphamide, procarbazine, prednisolone, etoposide, mitoxantrone, and bleomycin, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating older patients with previously untreated Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and toxicity of vinblastine, cyclophosphamide, procarbazine, prednisolone, etoposide, mitoxantrone, and bleomycin in older patients with Hodgkin's lymphoma.
* Determine whether the application of the Hasenclever prognostic index is valid in these patients at diagnosis.

OUTLINE: This is an open-label, multicenter study.

* Chemotherapy: Patients receive vinblastine IV and cyclophosphamide IV on day 1; oral procarbazine and oral prednisolone on days 1-5; oral etoposide on days 15-19; and mitoxantrone IV and bleomycin IV on day 15. Treatment repeats every 28 days, in the absence of disease progression or unacceptable toxicity, for a total of 3 courses in patients with early (stage IA or IIA) disease or 6 courses in patients with advanced (stage IB or IIB-IV) disease.
* Radiotherapy: Patients with early stage disease receive involved-field radiotherapy. Patients with advanced stage disease receive radiotherapy limited to sites of initial bulky disease or residual disease. Radiotherapy begins 4 weeks after the completion of chemotherapy.

Patients are followed monthly for 3 months, every 3 months for 6 months, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study within 36 months.

ELIGIBILITY:
Inclusion criteria:

Histologically confirmed classical Hodgkin Lymphoma (HL). No previous treatment for HL. Age ≥ 60. "Non fragile" patient (see Appendix 1) i.e. patient's mental and physical status must be sufficient to withstand the treatment described.

No concomitant neoplasia requiring treatment or known HIV infection. Written informed consent.

Exclusion criteria:

Nodular lymphocyte predominance Hodgkin Lymphoma (NLPHL) Age <60. Patient previously treated for HL. Known HIV infection or concomitant neoplasia. "Fragile patient" (see Appendix 1) or significant abnormality of another system (pulmonary, cardiac, renal, and hepatic) which is a contraindication to full dose chemotherapy.

Unable to give informed consent.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival by routine imaging | 6 month intervals

SECONDARY OUTCOMES:
Overall survival by routine imaging | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Proctor, MD, Study Chair — University of Newcastle Upon-Tyne; Helen H. Lucraft, MD, Study Director — Northern Centre for Cancer Treatment at Newcastle General Hospital; Katrina M. Wood, MD, Study Director — Sir James Spence Institute of Child Health at Royal Victoria Infirmary
Locations (54):
- Medizinische Universitaetsklinik I at the University of Cologne, Cologne, Germany
- United Kingdom (53):
  - Wansbeck General Hospital, Ashington, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Good Hope Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Cumberland Infirmary, Carlisle, England
  - Saint Richards Hospital, Chichester, England
  - University Hospital of North Durham, Durham, England
  - Queen Elizabeth Hospital, Gateshead-Tyne and Wear, England
  - Medway Maritime Hospital, Gillingham Kent, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Harrogate District Hospital, Harrogate, England
  - Hull Royal Infirmary, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Kettering General Hosptial, Kettering, Northants, England
  - Leeds General Infirmary, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - University College Hospital - London, London, England
  - Maidstone Hospital, Maidstone, England
  - Manchester Royal Infirmary, Manchester, England
  - Christie Hospital, Manchester, England
  - Trafford General Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - University of Newcastle-Upon-Tyne Northern Institute for Cancer Research, Newcastle upon Tyne, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - North Tyneside Hospital, North Shields, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Pembury Hospital, Royal Tunbridge Wells, Kent, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - University Hospital of North Staffordshire, Stoke-On-Trent Staffs, England
  - Sunderland Royal Hospital, Sunderland, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - West Cumberland Hospital, Whitehaven, England
  - Cancer Care Centre at York Hospital, York, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Monklands General Hospital, Airdrie, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Barnet General Hospital, Barnet, Hertfordshire

IPD SHARING:
Plan to Share IPD: No
No IPD were shared, nor will be, for this trial.